CLINICAL TRIAL: NCT05842798
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Following Intramuscular Administration of a Single Dose of TNM002 in Healthy Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of TNM002 in Chinese Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhuhai Trinomab Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: TNM002-P1-CH01
Record Dates: First submitted 2023-04-10; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: TNM002 35 μg/kg or placebo (Experimental): Eight subjects will be randomly assigned to receive either TNM002 35 μg/kg or placebo at a 3:1 ratio (i.e. 6 subjects receive TNM002 and 2 with placebo)
  Interventions: Drug: TNM002; Drug: Placebo
- Cohort 2: TNM002 100 μg/kg or placebo (Experimental): Eight subjects will be randomly assigned to receive either TNM002 100 μg/kg or placebo at a 3:1 ratio (i.e. 6 subjects receive TNM002 and 2 with placebo)
  Interventions: Drug: TNM002; Drug: Placebo
- Cohort 3：TNM002 250 μg/kg or placebo (Experimental): Eight subjects will be randomly assigned to receive either TNM002 250 μg/kg or placebo at a 3:1 ratio (i.e. 6 subjects receive TNM002 and 2 with placebo)
  Interventions: Drug: TNM002; Drug: Placebo

INTERVENTIONS:
Drug: TNM002 — TNM002, intramuscular injection
Drug: Placebo — Placebo, intramuscular injection

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics properties of TNM002 following a single intramuscular dose in Chinese healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, 18-55 years of age;
2. Body mass index (BMI) within 19.0-26.0 kg/m2;

Exclusion Criteria:

1. Any clinically significant chronic or acute medical condition that makes the volunteer unsuitable for participation;
2. Severe drug or excipient allergy, or history of hypersensitivity to other therapeutic mAbs;
3. History of alcohol or other substance abuse.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
AEs | Up to 105 days post dosing
  Incidence of AEs
Number of participants with clinically significant abnormality in physical examinations | Up to 105 days post dosing
  Clinically significant abnormality in general condition, skin, eyes/ears/nose/mouth/throat, neck/thyroid, chest/lungs, heart, vascular system, lymph nodes, abdomen, extremities, nervous systems/reflexes, musculoskeletal, spine
Change in Hematocrit (ratio) | Up to 105 days post dosing
  Measured by hematology test
Change in Haemoglobin (g/L) | Up to 105 days post dosing
  Measured by hematology test
Change in Platelet count (cells x 10^9/L) | Up to 105 days post dosing
  Measured by hematology test
Change in Red blood cell count (cells x 10^12/L) | Up to 105 days post dosing
  Measured by hematology test
Change in differential leukocyte count (cells x 10^9/L) | Up to 105 days post dosing
  Measured by hematology test
Change in Serum Alanine Aminotransferase (ALT) (U/L) | Up to 105 days post dosing
  Measured by serum chemistry
Change in Serum Aspartate Aminotransferase (AST) (U/L) | Up to 105 days post dosing
  Measured by serum chemistry
Change in Serum Albumin (g/L) | Up to 105 days post dosing
  Measured by serum chemistry
Change in Serum Alkaline Phosphatase (ALP) (U/L) | Up to 105 days post dosing
  Measured by serum chemistry
Change in Serum Total Bilirubin (umol/L) | Up to 105 days post dosing
  Measured by serum chemistry
Change in Serum Blood urea nitrogen (BUN) (mmol/L) | Up to 105 days post dosing
  Measured by serum chemistry
Change in Serum Creatinine (umol/L) | Up to 105 days post dosing
  Measured by serum chemistry
Change in Serum Calcium (mmol/L) | Up to 105 days post dosing
  Measured by serum chemistry
Change in Serum Chloride (mmol/L) | Up to 105 days post dosing
  Measured by serum chemistry
Change in Serum Cholesterol (mmol/L) | Up to 105 days post dosing
  Measured by serum chemistry
Change in Serum Creatine Kinase (U/L) | Up to 105 days post dosing
  Measured by serum chemistry
Change in Serum Glucose (mmol/L) | Up to 105 days post dosing
  Measured by serum chemistry
Change in Serum Lactate Dehydrogenase (U/L) | Up to 105 days post dosing
  Measured by serum chemistry
Change in Serum Phosphorus (mmol/L) | Up to 105 days post dosing
  Measured by serum chemistry
Change in Serum Potassium (mmol/L) | Up to 105 days post dosing
  Measured by serum chemistry
Change in Serum Total protein (g/L) | Up to 105 days post dosing
  Measured by serum chemistry
Change in Urine Bilirubin (U-BIL) | Up to 105 days post dosing
  Measured by Urinalysis
Change in Urine Glucose (GLU) (mg/dL) | Up to 105 days post dosing
  Measured by Urinalysis
Change in Urine erythrocytes (U-RBC) | Up to 105 days post dosing
  Measured by Urinalysis
Change in Urinary leukocyte (U-LEU) | Up to 105 days post dosing
  Measured by Urinalysis
Change in Urine nitrites (U-NIT) | Up to 105 days post dosing
  Measured by Urinalysis
Change in Urine protein (U-PRO) | Up to 105 days post dosing
  Measured by Urinalysis
Change in Urine specific gravity (U-SG) | Up to 105 days post dosing
  Measured by Urinalysis
Change in Urine urobilinogen (URO) | Up to 105 days post dosing
  Measured by Urinalysis
Change in Prothrombin time (sec) | Up to 105 days post dosing
  Measured by Blood Coagulation test
Change in Activated partial thromboplastin time (APTT)(sec) | Up to 105 days post dosing
  Measured by Blood Coagulation test
Change in fibrinogen (g/L) | Up to 105 days post dosing
  Measured by Blood Coagulation test
Change in international normalized ratio (INR | Up to 105 days post dosing
  Measured by Blood Coagulation test
Change in RR intervals (msec) | Up to 105 days post dosing
  Measured using a 12 Lead Electrocardiogram
Change in PR intervals (msec) | Up to 105 days post dosing
  Measured using a 12 Lead Electrocardiogram
Change in QRS duration (msec) | Up to 105 days post dosing
  Measured using a 12 Lead Electrocardiogram
Change in QT intervals (msec) | Up to 105 days post dosing
  Measured using a 12 Lead Electrocardiogram
Change in QTcB intervals (msec) | Up to 105 days post dosing
  Measured using a 12 Lead Electrocardiogram
Change in QTcF intervals (msec) | Up to 105 days post dosing
  Measured using a 12 Lead Electrocardiogram
Change in blood pressure (mmHg) | Up to 105 days post dosing
Change in pulse rate (bpm) | Up to 105 days post dosing
Change in body temperature (celsius) | Up to 105 days post dosing

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 105 days post dosing
  Estimated by non-compartmental analysis (NCA) with WinNonlin Version 7. 0 or above CL/F, Vz/F, MRT, λz, and %AUCex;
Time of maximum plasma concentration (Tmax) | Up to 105 days post dosing
  Estimated by non-compartmental analysis (NCA) with WinNonlin Version 7. 0 or above CL/F, Vz/F, MRT, λz, and %AUCex;
Terminal half-life (T1/2) | Up to 105 days post dosing
  Estimated by non-compartmental analysis (NCA) with WinNonlin Version 7. 0 or above CL/F, Vz/F, MRT, λz, and %AUCex;
Area under the plasma concentration-time curve from time-zero to the time of the last measurable concentration (AUC0-last) | Up to 105 days post dosing
  Estimated by non-compartmental analysis (NCA) with WinNonlin Version 7. 0 or above CL/F, Vz/F, MRT, λz, and %AUCex;
Area under the plasma concentration-time curve from time-zero extrapolated to infinite time (AUC0-inf) | Up to 105 days post dosing
  Estimated by non-compartmental analysis (NCA) with WinNonlin Version 7. 0 or above CL/F, Vz/F, MRT, λz, and %AUCex;
Apparent total body clearance (CL/F) | Up to 105 days post dosing
  Estimated by non-compartmental analysis (NCA) with WinNonlin Version 7. 0 or above CL/F, Vz/F, MRT, λz, and %AUCex;
Apparent volume of distribution (Vz/F) | Up to 105 days post dosing
  Estimated by non-compartmental analysis (NCA) with WinNonlin Version 7. 0 or above CL/F, Vz/F, MRT, λz, and %AUCex;
Anti-TNM002 antibodies | Up to 105 days post dosing
  The numbers of subjects who developed anti-TNM002 antibodies
Anti-TNM002 antibodies | Up to 105 days post dosing
  The percentages of subjects who developed anti-TNM002 antibodies

OTHER OUTCOMES:
Tetanus-antibody titer | Up to 105 days post dosing
  Geometric mean titers (GMTs) of tetanus-antibody titer in serum
Tetanus-antibody titer | Up to 105 days post dosing
  The percentage of subjects with a change of titer > 10 IU/L from the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Zhigang Liu, Principal Investigator — The Fifth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Fifth Affiliated Hospital Sun Yat-sen University, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in these articles after deidentification
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Academics who provide a methodologically sound proposal.